CLINICAL TRIAL: NCT04187768
Title: Immunological Profile Changes In Patients With Advanced Non-Small Cell Lung Cancer Undergoing Treatment With Checkpoint Inhibitor Monotherapy
Brief Title: Immunological Profile Changes In Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Nasser Hanna, Professor of Medicine, Tom and Julie Wood Family Foundation Professor of Lung Cancer Clinical Research, Indiana University
Other Study IDs: CTO-IUSCC-0701
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Non Small Cell Lung Cancer; Non Small Cell Lung Cancer Metastatic; Healthy
Keywords: Blood Donation; Lung Cancer; Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10 mL of blood will be collected at each time point
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Group: Healthy volunteers will donate a sample of blood to be used as controls
- NSCLC Group: Patients with advanced NSCLC will have blood collected prior to treatment and after completing 3 cycles of immune checkpoint therapy. . If a patient is noted to have progressive disease after 2 cycles of treatment, a sample will be collected after the 2nd cycle. If a patient is noted to have pseudoprogression (determined at the discretion of the treating physician), an additional sample may be collected after 3 cycles of therapy.

SUMMARY:
This is a blood collection study being conducted to better understand and describe the immunological blood profile changes in patients with advanced non small cell lung cancer undergoing treatment with checkpoint inhibitor therapy. Blood will be collected from healthy volunteers and patients with non small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent
2. Written informed consent and HIPAA authorization for release of personal health information.
3. Subjects with histologically and radiographically confirmed NSCLC.
4. Subjects must have stage IV disease or recurrent disease.
5. Subjects should be treatment naïve (systemic therapies) or have received prior chemotherapy in the first line setting. Prior radiation or surgery is permissible.
6. Subjects who are eligible to receive single agent immunotherapy must have documentation of a PD-L1 Tumor Proportion Score (TPS) of at least 1%.
7. Subjects with Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.

Exclusion Criteria:

1. Subjects with curable or potentially curable NSCLC.
2. Subjects should not have contraindications to treatment with immune checkpoint inhibitors per standard criteria.
3. Patients with targetable mutations eligible for treatment with molecularly targeted small molecule inhibitor therapy.
4. Subjects eligible for combination treatment with chemoimmunotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with advanced NSCLC and healthy volunteers with no diagnosis of cancer, known immunodeficiency or other serious chronic illness
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Mean change in myeloid derived suppressive cells (MDSCs) | baseline and cycle 3
  change in MDSCs before and after treatment
Mean change in B regulatory cells (Bregs) | baseline and cycle 3
  change in Bregs before and after treatment
Mean change in T regulatory cells (Tregs) before and after treatment | baseline and cycle 3
  change in Tregs before and after treatment

SECONDARY OUTCOMES:
Describe the programmed death-ligand 1 (PD-L1) expression profile on peripheral blood MDSCs, Bregs, and Tregs | baseline, cycle 3
Describe the programmed death-ligand 1 (PD1) expression profile on peripheral blood MDSCs, Bregs, and Tregs | baseline, cycle 3

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, MD, Principal Investigator — Indiana Unversity
Locations (1):
- Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana, United States